CLINICAL TRIAL: NCT06448182
Title: Precision Medicine Against Type 2 Diabetes: Genetic Prediction and Nutritional Intervention With Postbiotics to Modulate Microbiota.
Brief Title: Effect of a Postbiotic Intake on Glucose Control and Microbiota Composition of Type 2 Diabetic Subjects: a Randomized Controlled Trial.
Acronym: Diabet2Predict
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Biobizkaia (Unknown); Genbioma Aplicaciones S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIABET2PREDICT (2024.055)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Obesity; Postbiotic; Microbiota; Genetics; Randomized Controlled Trial; Supplementation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, parallel intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products (experimental and placebo), will be produced by an external producer, who will save the codes. None of the researchers involved in the study development or analyses will know the association until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotic group (Experimental): 1 postbiotic capsule daily in the morning during 12 weeks
  Interventions: Dietary Supplement: Postbiotic
- Placebo group (Placebo Comparator): 1 placebo capsule daily in the morning during 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Postbiotic — 1 capsule of postbiotic daily in the morning
  Arms: Postbiotic group
Dietary Supplement: Placebo — 1 capsule of placebo daily in the morning
  Arms: Placebo group

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effect of the administration of a postbiotic on glycemic control, insulin resistance and microbiota composition in subjects with type 2 diabetes.

The main questions it aims to answer are:

* Study the evolution of biochemical variables related to glycemic metabolism: basal glucose, basal insulin, glycemic variability through sensors, glycosylated hemoglobin (HbA1c), HOMA-IR index, C peptide.
* Perform a metagenomic analysis of intestinal microbiota in stool samples.
* Perform a metabolomics analysis on blood samples.
* Analyze the genetic profile in blood.
* Evaluate the evolution of biochemical variables related to lipid metabolism: total serum cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides.
* Assess the evolution of variables related to liver function: transaminases (ALT/AST).
* Analyze the evolution of the blood count.
* Evaluate the evolution of anthropometric variables (weight, height, waist and hip) and body composition.
* Analyze the evolution of blood pressure.
* Analyze eating and physical activity habits.
* Evaluate adherence to treatment and adverse events.
* Personalization on the use of postbiotics and other nutritional recommendations based on the genetic profile and the identification of patient clusters.

For this purpose, a randomized, double blind parallel study has been designed.

Target sample size is 158 subjects.

Participants will be allocated in two groups for 12 weeks:

* Experimental group (n=79): daily consumption of one postbiotic capsule.
* Placebo group (n=79): daily consumption of one placebo capsule.

Researchers will compare the consumption of a postbiotic supplement to a placebo.

Participants will visit nutritional intervention unit at week 0, week 2, week 10 and week 12 of the study.

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study will be interviewed by phone to verify that they meet the main inclusion criteria. Volunteers who meet the main inclusion criteria will be invited to an information and screening visit to resolve any doubts. Volunteers who agree to participate in the study will sign the informed consent and will be randomly allocated to one of the two arms of the study and will be provided with any required material.

During the intervention, volunteers will attend 4 Clinical investigation visits. The first one will be carried out on the first day of the study and the last one will take place at the end of the 12 weeks. In both visits anthropometric and body composition measurements, blood pressure, stool and blood samples, as well as data about dietary, physical activity and gastrointestinal symptoms will be taken. In the second and the third visits anthropometric, body composition, blood pressure and a blood sample will be taken. In the first and the third visits glucose monitoring sensor will be put and in the second and the fourth visits this glucosae monitoring sensor will be retired.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years.
* Subjects diagnosed with DM2: glycosylated hemoglobin (HbA1c) ≥6.5% and/or basal glucose ≥126 mg/dL. Debut time will not be taken into account.
* Body Mass Index (BMI) between 25 and 39.9 kg/m2.
* Treatment for DM2/stable lifestyle, as well as other treatments for other pathologies (stable at least 3 months prior to the start of the intervention).
* Stable baseline HbA1c or glucose value for at least 3 months before starting the intervention.
* No weight variations (± 5%) during the last 3 months.
* Subjects must be in general physical and psychological conditions that the researcher assesses in accordance with the objective of the study.
* Subjects must be able to understand and be willing to sign the informed consent, and must comply with all study procedures and requirements.

Exclusion Criteria:

* Subjects who have received oral antibiotic treatment in the 45 days prior to the start of the study.
* Patients who have started hypoglycemic treatment, especially in the 3 months prior to inclusion. Insulin treatment.
* Severe untreated dyslipidemia, hypertension or hypothyroidism, or treated for less than 3 months.
* Presence of relevant functional or structural anomalies of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory diseases or malabsorption.
* Subjects who have undergone surgical interventions of the digestive system with permanent consequences (for example, gastroduodenostomy).
* Suffer from any type of cancer or be undergoing treatment for it, or a period of less than 5 years since its eradication.
* Subjects who work rotating shifts that include night shifts.
* Presence of some type of psychological impediment such as depressive pathology, anxiety, untreated bipolar disorder. They will be able to participate if they have the disease but with stable treatment for at least 3 months prior to the start of the trial.
* Have an allergy or intolerance to any food or food group that is likely to manifest during the study.
* Be on a special diet during the 3 months prior to the start of the study, except for treatment for DM2, in this case, the lifestyle/diet will have to be stable in the 3 months prior to the start of the study.
* Weight variations (± 5%) during the last 3 months.
* Suffer from eating disorders or present restrictive behaviors in their diet. Score on the EAT-26 questionnaire equal to or greater than 20.
* Subjects who have undergone surgical treatment for obesity.
* Be pregnant or breastfeeding.
* Present alcohol abuse (more than 14 units/day in women and 20 units/day in men) and/or drugs.
* Show poor collaboration or have difficulties to follow the study procedures.
* Take some type of nutritional supplementation that can affect blood glucose and/or the microbiota. If they take it, in order to be included in the study, they will have to stop the supplement, with a washout period of at least 14 days before starting the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood glycated hemoglobin (HbA1c) concentration | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood glycated hemoglobin will be analysed in total blood and reported in % and in mmol/mol.

SECONDARY OUTCOMES:
Change from baseline in blood glucose | Clinical Investigation Days 1 (week 0), 2 (week 2), 3 (week 10) and 4 (week 12).
  Blood will be extracted at fasting state and glucose levels will be determined by autoanalyzer Pentra-C200.
Change from baseline in blood insulin | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and insulin levels will be determined by ELISA.
Continuous glucose levels | Clinical Investigation Day 1 (week 0) to Clinical Investigation Day 2 (week 2) and Clinical Investigation Day 3 (week 10) to Clinical Investigation Day 4 (week 12).
  Continuous glucose levels will be controlled with FreeStyle Libre Pro (Abbott) glucose monitoring sensor.
Change from baseline in blood Peptide C | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and peptido C levels will be determined by ELISA.
Change from baseline in hemogram | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and hemogram profile will be determined by autoanalyzer Pentra-C60.
Change from baseline in fecal microbiota | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Fecal microbiota of participants will be analyzed by bacterial 16S gene sequencing technology.
Blood genetic profile | Clinical investigation day 1
  Genetic profile will be analysed in blood of participants.
Change from baseline in blood total cholesterol | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and Total cholesterol levels of participants will be analysed by autoanalyzer Pentra-C200.
Change from baseline in blood HDL cholesterol | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and HDL cholesterol levels of participants will be analysed by autoanalyzer Pentra-C200.
Change from baseline in blood LDL cholesterol | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  LDL cholesterol levels of participants will be calculted by Friedewald equation.
Change from baseline in blood tryglicerides | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and trygliceride levels of participants will be analysed by autoanalyzer Pentra-C200.
Change from baseline in blood lactate | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and lactate levels of participants will be analysed by autoanalyzer Pentra-C200.
Change from baseline in blood alanine aminotransferase (ALT) | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and ALT levels of participants will be analysed by autoanalyzer Pentra-C200.
Change from baseline in blood aspartate aminotransferase (AST) | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Blood will be extracted at fasting state and AST levels of participants will be analysed by autoanalyzer Pentra-C200.
Change from baseline in body weight | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Weight of participants will be measured by bioimpedance and reported in kg.
Height | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Height of participants will be measured by stadiometer and reported in m.
Change from baseline in body mass index | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Body mass index will be calculated as follows: weight (kilograms)/ height (cm)2.
Change from baseline in body fat percentage | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Body fat of participants will be analyzed by bioimpedance and reported in percentage and kilograms.
Change from baseline in body muscle mass | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Body muscle mass of participants will be analyzed by bioimpedance and reported in kilograms.
Change from baseline in body lean mass | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Body leen mass of participants will be analyzed by bioimpedance and reported in kilograms.
Change from baseline in body water mass | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Body water mass of participants will be analyzed by bioimpedance and reported in kilograms.
Change from baseline in body bone mass | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Body bone mass of participants will be analyzed by bioimpedance and reported in kilograms.
Change from baseline in waist circumference | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change from baseline in hip circumference | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change from baseline in systolic blood pressure | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change from baseline in diastolic blood pressure | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change from baseline in heart rate | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change from baseline in gastrointestinal symptoms | Clinical investigation day 1 (week 0), 2 (week 2), 3 (week 10) and 4 (week 12).
  Gastrointestinal symptoms will be registrated through Gastrointestinal Symptoms Rating Scale questionnaire, which is a questionnaire of 15 items. The questionnaire has a seven-point graded likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Change from baseline in physical activity | Clinical investigation day 1 (week 0) and 4 (week 12).
  Physical activity will be evaluated by the reduced version of the International Physical Activity Questionnaire, which estimates the total physical activity in MET-min/week, time spent sitting and classifies subjects based on their physical activity.
Change from baseline in global dietary intake | Clinical Investigation Day 1 (week 0) and Clinical Investigation Day 4 (week 12).
  Global dietary intake (energy, macronutrients and micronutrients) will be analysed by food frequency questionnaire.
Change from baseline in adherence to capsule consumption | Clinical investigation day 1 (week 0), 2 (week 2), 3 (week 10) and 4 (week 12).
  Adherence will be assessed using the capsule consumption record form.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro González-Muniesa, PhD, Principal Investigator — Nutrition Research Centre
Locations (3):
- Spain (3):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Nutrition Research Centre, University of Navarra, Pamplona, Navarre
  - IIS Biobizkaia, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: No